CLINICAL TRIAL: NCT04395105
Title: High Versus Low Dose Dexamethasone for the Treatment of COVID-19 Related ARDS: a Multicenter and Randomized Open-label Clinical Trial
Brief Title: Dexamethasone for COVID-19 Related ARDS: a Multicenter, Randomized Clinical Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low rate of recruitment
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Principal Investigator, Pablo Oscar Rodriguez, Pulmonary and Critical Care Coordinator, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1264
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Distress Syndrome, Adult; Covid-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose Dexamethasone (Experimental): Intravenous Dexamethasone 16 mg qd from day 1 to 5 followed by 8 mg qd from day 6 to 10
  Interventions: Drug: High-Dose Dexamethasone
- Usual care - low dose Dexamethasone (No Intervention): Intravenous Dexamethasone 6 mg qd for 10 days based on RECOVERY trial

INTERVENTIONS:
Drug: High-Dose Dexamethasone — IV Dexamethasone administered once daily: 16 mg from day 1 to 5 and 8 mg from day 6 to 10
  Other Names: Corticosteroid
  Arms: High dose Dexamethasone

SUMMARY:
There is compelling data indicating that there is an excessive inflammatory response in some patients with COVID-19 leading them to develop ARDS that can be severe with a very poor prognosis. Many of these patients require very long mechanical ventilation times to survive, which have led to the collapse of the health system in some regions of the world. The current evidence for the treatment of these severe forms is inconsistent and most scientific societies and governmental or international organizations recommend evaluating treatments with randomized clinical trials. Corticosteroids, being non-specific anti-inflammatory drugs, could shorten the duration of respiratory failure and improve the prognosis. Due to the lack of solid data available regarding this serious disease, our objective is to randomly evaluate the efficacy and safety of the use of dexamethasone, a parenteral corticosteroid approved in Argentina, in patients with ARDS with confirmed respiratory infection due to SARS-CoV-2 (COVID-19).

After RECOVERY trial prepublication, low dose (6 mg QD for 10 days) dexamethasone was recommended as the usual care treatment for severe COVID-19. At this time only 3 patients had been included in the trial. Thus, we updated our recommendations for centers and decided to compare two different doses of this glucocorticoid for the treatment of ADRS due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* ARDS according to Berlin's definition
* PCR confirmed COVID-19
* Length of mechanical ventilation less or equal to 72 hours

Exclusion Criteria:

* Pregnancy or breast-feeding women
* Terminal illness with very poor prognosis according to the investigator judgement
* Therapeutic limitation
* Known immunocompromised condition
* Chronic use of systemic corticosteroids
* Participation in another randomized crinical trial
* More than 5 days of treatment of low dose dexamethasone for COVID-19
* Abscence of informed consent
* Active participation in other randomized clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days at 28 days | 28 days after randomization
  Days without ventilator support in the first 28 days following randomization
Time to successful discontinuation from mechanical ventilation | 28 days after randomization
  Time to event (successful discontinuation from mechanical ventilation)

SECONDARY OUTCOMES:
28-days mortality | 28 days after randomization
  Dead rate within 28 days of randomization
Rate of nosocomial infections | 28 days after randomization
  Rate of ventilator associated pneumonia, blood stream infection, urinary tract infection or candidemia in the first 28 days following randomization
SOFA variation | 10 days after randomization
  Variation in SOFA over the first 10 days after randomization
Use of prone position | 10 days after randomization
  Cumulative hours spent on prone position
Delirium | 28 days after randomization
  Frequency of delirium at ICU discharge
Muscle weakness | 28 days after randomization
  mMRC score at ICU discharge
90-day mortality | 90 days after randomization
  Death rate within 90 days of randomization
Peak daily blood glucose | 10 days after randomization
  Interaction between treatment and daily change in glucose

CONTACTS AND LOCATIONS:
Overall Officials: Pablo O Rodriguez, MD, Principal Investigator — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno; Luis P Maskin, MD, Principal Investigator — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Locations (4):
- Argentina (4):
  - Clínica Bazterrica, Buenos Aires
  - Hospital Universitario Sede Pombo - IUC CEMIC, Buenos Aires
  - Sanatorio Sagrado Corazon, Buenos Aires
  - Hospital Universitario Sede Saaveda - IUC CEMIC, CABA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maskin LP, Olarte GL, Palizas F Jr, Velo AE, Lurbet MF, Bonelli I, Baredes ND, Rodriguez PO. High dose dexamethasone treatment for Acute Respiratory Distress Syndrome secondary to COVID-19: a structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Aug 26;21(1):743. doi: 10.1186/s13063-020-04646-y. PMID 32843098
- See also: Protocol publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7447582